CLINICAL TRIAL: NCT05695729
Title: Effects of Upper Body Plyometrics Versus Conventional Exercises on Speed, Strength and Injury Prevention in Bowlers.
Brief Title: Effects of Plyometrics Versus Conventional Exercises on Speed, Strength, and Injury Prevention in Bowlers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC/01403 Ibtahaj ul Islam
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Sports Injury; Sports Physical Therapy
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLYOMETRIC EXERCISE PROGRAM GROUP (Experimental): The Plyometric exercise group will receive 8 weeks of upper body plyometric exercise protocol. The session will last for 60 minutes 3 times per week.
  Exercises will be done according to FIIT protocol.
  Interventions: Other: PLYOMETRIC EXERCISE PROGRAM
- CONVENTIONAL EXERCISE PROGRAM GROUP (Active Comparator): The conventional group will receive 8 weeks of upper body strength exercise protocol. The session will last for 60 minutes 3 times per week.
  Exercises will be done according to FIIT protocol.
  Interventions: Other: CONVENTIONAL EXERCISE PROGRAM

INTERVENTIONS:
Other: PLYOMETRIC EXERCISE PROGRAM — This group will perform following exercises in first four weeks. Reverse overhead throw Rotational wall throws Overhead medicine ball Chest passes Resistance tubing 90-90 external rotation
  Frequency
  * Rest between Exercises-: 60-120 Seconds
  * Rest between Set of Exercise-: 45-60 Seconds after four weeks rest between exercise and rest between set of exercise will be reduced:
  * Rest between Exercises-: 45-60 Seconds
  * Rest between Set of Exercise-: 20-30 Seconds
  Tools used:
  Medicine Ball, Resistance band
  Arms: PLYOMETRIC EXERCISE PROGRAM GROUP
Other: CONVENTIONAL EXERCISE PROGRAM — This group will perform following exercise through out the session with different frequencies after 4 weeks Bench presses Triceps kickbacks bicep curls Overhead presses Push-ups
  Frequency:
  Rest between Exercises-: 60-120 Seconds Rest between Set of Exercise-: 45-60 Seconds
  After 4 weeks the frequency will be:
  Rest between Exercises-: 45-60 Seconds Rest between Set of Exercise-: 20-30 Seconds
  Arms: CONVENTIONAL EXERCISE PROGRAM GROUP

SUMMARY:
To compare the effects of upper body plyometric versus conventional exercises on speed, strength, and injury prevention in bowlers

DETAILED DESCRIPTION:
Bowling action is a highly skilled activity acquired over the year. A bowler needs speed and strength to challenge the batsman but the conventional protocols they follow for the speed and strength are not specific to their bowling actions. Bowling can result in different types of upper extremity injuries, such as rotator cuff sprains, impingement and stress fractures. There are many injury prevention programs such as electrostimulation training, resistance training, and plyometric training that can be used to treat upper limb injuries and improve maximal strength.

Plyometric training can be done by overhead athletes to improve the effectiveness of throwing activity and to strengthen the rotator cuff muscles to prevent shoulder injury from overhead throwing activity.

This study aims to evaluate the effectiveness of upper limb plyometric exercises on speed, strength and injury prevention in comparison with conventional exercises.

ELIGIBILITY:
Inclusion Criteria:

* Players bowling for at least one year
* Bowlers age 18 to 35 years

Exclusion Criteria:

* Any acute or chronic musculoskeletal injuries
* Any surgery in 6 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Strength | 8 weeks
  Seated power throw (medicine ball) will be used to assess strength and explosive power of the upper body. The athlete sits on the floor with his legs fully extended, feet 24 inches (~60 cm) apart and with the back against a wall. The ball is held with the hands on the side and slightly behind the centre and back against the centre of the chest. The forearms are positioned parallel to the ground. The athlete throws the medicine ball vigorously as far straight forward as he can while maintaining the back against the wall. The distance thrown is recorded.
Speed | 8 weeks
  Speed gun will be used to assess the speed of a ball thrown by a bowler from one end of the pitch to another end.

SECONDARY OUTCOMES:
Injury Prevention | 8 weeks
  DASH questionnaire (Reliability: ICC = 0.96, Validity: r > 0.70) It is a 30-item questionnaire that look the ability of a patient to perform certain upper extremity activities. This is a self-report questionnaire that patient can rate difficulty and interference with daily life on a 5-point Likert chart.

CONTACTS AND LOCATIONS:
Overall Officials: Saad Rauf, Ph.D*, Principal Investigator — Riphah International University
Locations (1):
- Ayub Stadium, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: No